CLINICAL TRIAL: NCT00002696
Title: MULTIMODALITY TREATMENT STRATEGY FOR STAGE III BREAST CANCER
Brief Title: Combination Chemotherapy in Treating Women With Stage III Breast Cancer
Status: Suspended | Phase: Phase 3 | Type: Interventional
Sponsor: Grupo Oncologico Cooperativo del Sur (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: GOCS-08-BR-95-III; CDR0000064471 (Registry Identifier: PDQ (Physician Data Query)); NCI-F95-0036
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2008-04

CONDITIONS: Breast Cancer
Keywords: stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — CAF protocol; CMF regimen; Cyclophosphamide; Doxorubicin; Fluorouracil; Methotrexate; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Radiotherapy

INTERVENTIONS:
Drug: CAF regimen
Drug: CMF regimen
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: fluorouracil
Drug: methotrexate
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Randomized phase III trial to compare cyclophosphamide, doxorubicin, and fluorouracil with cyclophosphamide, methotrexate, and fluorouracil in treating women with stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the response in women with stage III breast cancer treated with neoadjuvant fluorouracil, doxorubicin, and cyclophosphamide (FAC) vs cyclophosphamide, methotrexate, and fluorouracil (CMF).
* Compare the rates of conservative surgical resectability and locoregional control in patients treated with these neoadjuvant therapy regimens.
* Compare the disease-free and overall survival of patients treated with these regimens.
* Compare the toxic effects of these regimens in these patients.
* Compare the compliance of patients treated with these regimens.
* Assess the cosmetic results in patients treated with conservative surgery.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center.

* Arm I: Patients receive fluorouracil (5-FU) IV on days 1 and 8 and doxorubicin IV and cyclophosphamide (CTX) IV on day 1 (FAC). Treatment continues every 3 weeks for 3 courses in the absence of disease progression.
* Arm II: Patients receive CTX IV, methotrexate IV, and 5-FU IV on days 1 and 8 (CMF). Treatment continues every 4 weeks for 3 courses in the absence of disease progression.

Patients on both arms with resectable disease after the third course of chemotherapy undergo quadrantectomy with axillary node dissection (preferred) or modified radical mastectomy, followed by 6 additional courses of chemotherapy on the arm to which they were randomized initially. Those patients without distant metastasis undergo locoregional radiotherapy beginning concurrently with the initiation of postoperative chemotherapy. Patients on both arms with unresectable disease after the initial 3 courses of chemotherapy undergo locoregional radiotherapy and then surgical resection (if feasible).

Quality of life is assessed at baseline and then monthly thereafter.

Patients are followed every 3-4 months for 2 years, every 4-6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: Not specified

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage III breast cancer
* Measurable disease
* No inflammatory breast cancer
* No synchronous bilateral breast cancer
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 21 to 75

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* ECOG 0-1 OR
* Zubrod 0-1

Life expectancy:

* More than 12 weeks

Hematopoietic:

* WBC greater than 4,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin less than 1.25 times upper limit of normal (ULN)
* AST less than 1.25 times ULN

Renal:

* Creatinine clearance greater than 70 mL/min

Cardiovascular:

* No angina pectoris
* No significant arrhythmia requiring therapy
* No bilateral bundle branch block
* No congestive heart failure
* No myocardial infarction

Other:

* No medical or psychiatric disease that would preclude study therapy
* No other malignancy except adequately treated nonmelanomatous skin cancer or carcinoma in situ of the cervix
* Not pregnant

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy

Surgery:

* No prior surgery except incisional biopsy or fine-needle aspiration

Other:

* No prior systemic therapy
* No concurrent caffeine or alcohol

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1995-10

CONTACTS AND LOCATIONS:
Overall Officials: Bernardo A. Leone, MD, Study Chair — Unidad Oncologica Del Neuquen
Locations (7):
- Argentina (7):
  - Policlinica Privada Instituto De Medicina Nuclear, Bahía Blanca, Buenos Aires
  - Consultorio Oncologico Privado, Mar del Plata, Buenos Aires
  - Centro De Oncologia y Terapia Radiante, Santa Rosa, La Pampa Province
  - Unidad Oncologica Del Comahue, Neuquén, Neuquén Province
  - Consultorio Oncologico Privado, Río Gallegos
  - Centro Oncologico Del Litoral, Santa Fe
  - Centro Oncologico Tres Arroyos, Tres Arroyos